CLINICAL TRIAL: NCT00536081
Title: Primary G-CSF Prophylaxis During the First Two Cycles Only or Throughout All Chemotherapy Cycles in Breast Cancer Patients at Risk of Febrile Neutropenia
Brief Title: Various G-CSF Regimens to Prevent Infection During Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, V.C.G. Tjan-Heijnen, Prof. dr., Academisch Ziekenhuis Maastricht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2-2-6 STUDY; ZonMw ID 80-82310-98-08006 (Other Grant/Funding Number: Stichting ZonMW); EudraCT number 2007-005402-53 (Other: Centrale Commissie Mensgebonden Onderzoek CCMO)
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Chemotherapy; Febrile Neutropenia
Keywords: Breast cancer; Adjuvant; Advanced; Chemotherapy; G-CSF; Pegfilgrastim; Prevention; Febrile neutropenia
MeSH Terms: conditions — Breast Neoplasms; Febrile Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Pegfilgrastim during all 6 cycles of chemotherapy
  Interventions: Drug: pegfilgrastim
- B (Experimental): Pegfilgrastim during the first two cycles of chemotherapy
  Interventions: Drug: pegfilgrastim

INTERVENTIONS:
Drug: pegfilgrastim — 6 mg s.c. 24-36 h post-chemotherapy

SUMMARY:
The purpose of this study is to prevent chemotherapy-related febrile neutropenia, prophylaxis with antibiotics and granulocyte colony-stimulating factor (G-CSF) have proven efficacious [1-3]. G-CSF has only few side effects, but is expensive. In 2006, updated G-CSF guidelines conclude that primary G-CSF prophylaxis has clinical benefits for and should be offered to patients at a more than 20% risk of febrile neutropenia.

Based on many positive and few negative trials, one can consider the use of taxanes as standard of care in the adjuvant setting in node-positive breast cancer. Taxanes (with or without anthracyclines) have an increased risk for febrile neutropenia.

The updated guidelines and changes in daily clinical practice will have a significant impact on the investigators health care resources. There is a higher risk of febrile neutropenia for the first chemotherapy cycle compared to subsequent cycles in small cell lung cancer patients. Also in advanced breast cancer the majority of first observed episodes of febrile neutropenia occur in the initial chemotherapy cycles Irrespective of tumour type or chemotherapy regimen, the risk of febrile neutropenia is highest during the first two cycles of chemotherapy. Thereafter, the risk rapidly declines, and the benefit of G-CSF largely seems to disappear.

So, in order to improve the cost-effective administration of primary G-CSF prophylaxis, it is justified to assess whether G-CSF prophylaxis can be limited to the first two chemotherapy cycles as compared to the current practice of continuous G-CSF prophylaxis.

DETAILED DESCRIPTION:
1. Febrile neutropenia Febrile neutropenia is a serious side effect of cancer treatment. Febrile neutropenia predisposes to serious and sometimes life-threatening infections. Given the seriousness, the majority of febrile neutropenia patients are admitted to hospital for treatment with intravenous antibiotics. Thus, chemotherapy-induced febrile neutropenia can result in death, increased hospitalisations and intravenous antibiotic use. In addition, it can lead to significant chemotherapy dose modifications, which may theoretically be of concern for treatments with curative intent. Clearly, prevention of chemotherapy-induced febrile neutropenia is a medical priority.

2 Prophylaxis of febrile neutropenia To prevent chemotherapy-related febrile neutropenia, prophylaxis with antibiotics and granulocyte colony-stimulating factor (G-CSF) have proven efficacious [1-3]. The use of the G-CSF was shown to shorten the duration of neutropenia, resulting in reduction of the incidence of febrile neutropenia, hospitalisation and use of intravenous therapeutic antibiotics by approximately 50%. .Antibiotics may, however, lead to emergence of microbial resistance. G-CSF has only few side effects, but is expensive. Previous guidelines recommended primary G-CSF prophylaxis to prevent febrile neutropenia, but only for patients at substantial risk of febrile neutropenia (more than 40%). In 2006, updated G-CSF guidelines conclude that primary G-CSF prophylaxis has clinical benefits for and should be offered to patients at a more than 20% risk of febrile neutropenia.

Most of the recent EORTC-reviewed evidence indicate that primary and secondary G-CSF prophylaxis had no significant impact on survival, despite the fact that G-CSF prophylaxis enabled to maintain chemotherapy dose and dose intensity. In the GEICAM 9805 study, primary G-CSF support did not lead to improved median dose intensity or cumulative dose when compared to secondary G-CSF prophylaxis, although the percentage of patients who completed six cycles of therapy increased significantly.

3. Developments in the adjuvant treatment of breast cancer After the introduction of taxanes in the treatment of advanced breast cancer in the late nineties, these agents have now also been introduced in the (neo) adjuvant setting. Many adjuvant trials with a positive outcome have recently been reported.

Based on the available data with many positive and few negative trials, one can consider the use of taxanes as standard of care in the adjuvant setting in node-positive breast cancer, although the preferred schedule, concurrent or sequential, with or without dose-densification, needs to be clarified from ongoing trials.

Martin et al. report on the results of a randomized adjuvant trial comparing TAC with FAC for high-risk N0 breast cancer patients, the GEICAM 9805 trial. Comparisons are reported for toxicity and quality of life. Only secondary G-CSF prophylaxis was allowed or even mandatory after an episode of febrile neutropenia. After a protocol amendment, patients in the TAC arm received primary G-CSF prophylaxis. So, in addition to the upfront planned comparison of TAC versus FAC, the unplanned comparison of TAC-pre versus TAC-post amendment is reported. This comparison is very interesting, as it is to our knowledge the first comparison of primary versus secondary G-CSF prophylaxis ever reported. The use of primary G-CSF prophylaxis significantly reduced the incidence of febrile neutropenia associated with TAC chemotherapy. The percentage of patients with febrile neutropenia in one or more cycles was 24.6% and 6.5% in TAC-pre and TAC-post, respectively. Of note, in the TAC-pre group 71.1% of patients had received secondary G-CSF prophylaxis during on average 4 cycles of treatment. In the FAC group, only 2.3% of patients had febrile neutropenia as per protocol definition.

So, the combined use of anthracyclines and taxanes come with considerable increased risk of febrile neutropenia. Perez concluded in an editorial in the New England Journal of Medicine that on the basis of the available data, one can consider TAC (docetaxel, adriamycin, cyclophosphamide) to be a standard of care, as is the dose-dense regimen of doxorubicin and cyclophosphamide followed by paclitaxel, for patients with node-positive breast cancer. With this regimen, prophylactic growth-factor support is necessary to ameliorate myelosuppression and febrile neutropenia.

4. Consequences for health care costs We have recently reported that, even for patients with a considerable risk of febrile neutropenia, primary G-CSF prophylaxis comes with considerable extra costs in the Netherlands: on average € 5,123 per patient who have a baseline risk of febrile neutropenia of 32%. The updated guidelines and changes in daily clinical practice will have a significant impact on our health care resources. In the Netherlands several thousands of patients with many tumour types will require primary G-CSF prophylaxis, leading to an cost increase of at least € 10-20 million per year.

5. Rationale for the present study It has been demonstrated that there is a higher risk of febrile neutropenia for the first chemotherapy cycle compared to subsequent cycles in small cell lung cancer patients. Also in advanced breast cancer the majority of first observed episodes of febrile neutropenia occur in the initial chemotherapy cycles. With primary G-CSF prophylaxis the absolute neutrophil count nadir is less deep and of shorter duration in later cycles compared to the first cycle. This may suggests that there may be a priming effect of G-CSF to subsequent cycles, emphasizing that administration of G-CSF early in the course of treatment might be important.

So, irrespective of tumour type or chemotherapy regimen, the risk of febrile neutropenia is highest during the first two cycles of chemotherapy. Thereafter, the risk rapidly declines, and the benefit of G-CSF largely seems to disappear.

So, in order to improve the cost-effective administration of primary G-CSF prophylaxis, it is justified to assess whether G-CSF prophylaxis can be limited to the first two chemotherapy cycles as compared to the current practice of continuous G-CSF prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients ≥18 years.
* Indication for 3-weekly chemotherapy.
* Considered fit enough to receive chemotherapy, with adequate renal and hepatic function.
* Planned a chemotherapy regime in adjuvant, neo-adjuvant, advanced setting with an increased risk of febrile neutropenia, i.e.:
* Regimes with >20% risk of febrile neutropenia:

  * e.g. TAC (docetaxel, adriamycin, cyclophosphamide)
  * AT (adriamycin, docetaxel)
* Regimes with 10-20% risk of febrile neutropenia (e.g. AC, doxorubicin and vinorelbine, or docetaxel monotherapy) in the presence of ≥1 patient risk factor (>65 yrs, extensive bone marrow involvement or prior extensive radiotherapy on bone tissue
* Prior chemotherapy
* ECOG performance status of 2 or more, grade 2 or higher liver function abnormalities).
* That is, patients starting with docetaxel as second part of FEC-D are eligible for the last 3 docetaxel cycles, if there is an increased risk of febrile neutropenia, e.g. by elderly age.
* Able to comply with the protocol.
* Written informed consent obtained prior to any study specific screening.

Exclusion Criteria:

* Active uncontrolled infection.
* Inadequate renal or hepatic function.
* Any evidence or history of hypersensitivity or other contraindications to G-CSF medication.
* Not recovered from acute toxicities of prior therapies.
* Absolute neutrophil count (ANC) <1.5 x 109/l, not caused by bone marrow involvement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
number of febrile neutropenia episodes costs per treatment arm | 18 weeks (all chemotherapy cycles)

SECONDARY OUTCOMES:
Febrile neutropenia rates per cycle number. Other haematological and non-haematological toxicities. Number of chemotherapy cycles delivered. Dose and dose-intensity of chemotherapy. Disease progression. Number of toxic deaths per treatment arm. | 18 weeks (all chemotherapy cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Vivianne CG Tjan-Heijnen, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (21):
- Netherlands (21):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Ziekenhuis Rijnstate, Alysis, Arnhem
  - Wilhelmina Ziekenhuis, Assen
  - Slingeland Ziekenhuis, Doetinchem
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Ziekenhuis St. Jansdal, Harderwijk
  - Elkerliek Ziekenhuis, Helmond
  - Diaconessenhuis Leiden, Leiden
  - Leids Universitair Medisch Centrum, Leiden
  - University Hospital Maastricht, Maastricht
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - UMC St. Radboud, Nijmegen
  - Erasmus MC - Daniel den Hoed, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Orbis Medisch Centrum, Sittard
  - Mesos Medisch Centrum, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Ziekenhuis Zevenaar, Alysis, Zevenaar

REFERENCES:
- [Derived] Aarts MJ, Grutters JP, Peters FP, Mandigers CM, Dercksen MW, Stouthard JM, Nortier HJ, van Laarhoven HW, van Warmerdam LJ, van de Wouw AJ, Jacobs EM, Mattijssen V, van der Rijt CC, Smilde TJ, van der Velden AW, Temizkan M, Batman E, Muller EW, van Gastel SM, Joore MA, Borm GF, Tjan-Heijnen VC. Cost effectiveness of primary pegfilgrastim prophylaxis in patients with breast cancer at risk of febrile neutropenia. J Clin Oncol. 2013 Dec 1;31(34):4283-9. doi: 10.1200/JCO.2012.48.3644. Epub 2013 Oct 28. PMID 24166522
- See also: University Hospital Maastricht — http://www.azm.nl